CLINICAL TRIAL: NCT03092739
Title: A Non-Interventional Multinational Study to Assess PD-L1 Expression in Cytological Versus Histological Non-Small Cell or Small Cell Lung Cancer Specimens
Brief Title: A Study to Assess Programmed Death Ligand-1 (PD-L1) Expression in Cytological Versus Histological Lung Cancer Specimens
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO29978
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin fixed, paraffin embedded tumor tissue; formalin fixed paraffin embedded cytological samples (cell blocks) from the same participant will be retained until end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cytological and Histological Samples: Cytological and histological specimens that meet the eligibility criteria will be analyzed only from those participants who have consented to biomarker research, according to local regulations and ethical guidelines. Cytological samples may originate from fine needle aspirations. Pleural effusions or bronchial cytology samples (brushings and washings) may be allowed. Histological samples may originate from core needle biopsies, bronchial biopsies (thoracoscopy or mediastinoscopy) or surgical tissue resections.
  Interventions: Diagnostic Test: PD-L1 Immunocytochemistry (ICC); Diagnostic Test: PD-L1 Immunohistochemistry (IHC)

INTERVENTIONS:
Diagnostic Test: PD-L1 Immunocytochemistry (ICC) — PD-L1 expression in the cytological specimens will be assessed using different antibodies.
Diagnostic Test: PD-L1 Immunohistochemistry (IHC) — PD-L1 expression in the histological specimens will be assessed using different antibodies.

SUMMARY:
The primary purpose of this non-interventional, multinational study is to assess the feasibility of assessing PD-L1 protein expression on cytological samples as a surrogate for histological samples obtained from participants with any stage of non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Samples must have been collected in a manner that is compliant with local ethics committee guidance
* Samples must originate from participants diagnosed with NSCLC or SCLC
* Participants must have a pair of at least one cytological and one histological specimen that: Both originate from inside the thorax or from the same ex-thoracic site; Are confirmed to have been collected within a window no more than 6 weeks apart from each other; and are in compliance with the protocol defined sample requirements for histological and cytological specimens

Exclusion Criteria:

* Immune checkpoint inhibitor therapy from 4 weeks prior to collection of the first tumor sample until collection of the second matched sample

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with any stage of NSCLC or SCLC who have cytological and histological samples available.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Total Tumor Cells (TC) That Display Discernible PD-L1 Staining of any Intensity in Histological and Cytological Samples As Assessed Using PD-L1 IHC/ICC Assay | approximately 12 months
Percentage of Total TC Within ten High-Power Fields (HPF) That Display Discernible PD-L1 Staining of any Intensity in Histological and Cytological Samples As Assessed Using PD-L1 IHC/ICC Assay | approximately 12 months
Percentage of Total Tumor Area That Contain Tumor-Infiltrating Immune Cells of any Discernible PD-L1 Staining of any Intensity in Histological Samples As Assessed Using PD-L1 IHC Assay | approximately 12 months
Percentage of Total Immune Cells That Display Discernible PD-L1 Staining of any Intensity in Cytological Samples As Assessed Using PD-L1 ICC Assay | approximately 12 months
Percentage of Total Immune Cells Within ten HPF That Display Discernible PD-L1 Staining of any Intensity in Histological and Cytological Samples As Assessed Using PD-L1 IHC/ICC Assay | approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Vseobecna fakultni nemocnice v Praze; I. klinika tuberkulozy a respiracnich nemoci, Prague, Czechia
- Universitätsklinikum Göttingen, Institut für Pathologie, Göttingen, Germany
- Instytut Gruźlicy i Chorób Płuc, I Klinika Chorób Płuc, Warsaw, Poland
- Spain (3):
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Anatomía Patológica, A Coruña, LA Coruña
  - Hospital Universitario La Paz; Servicio de Anatomia Patologica, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- C. INTEGRAL ONC. CLARA CAMPAL; Servicio Anatomia Patologica, Madrid
- Universitätsspital Basel; Pathologie, Basel, Switzerland
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No